CLINICAL TRIAL: NCT05767645
Title: Mistral Percutaneous Tricuspid Valve Durable Repair Pivotal Study
Acronym: TRIBUTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mitralix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-1048
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mistral device (Experimental): The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Tricuspid Regurgitation (TR).
  The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.
  Interventions: Device: Mistral Procedure

INTERVENTIONS:
Device: Mistral Procedure — The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Tricuspid Regurgitation (TR).
  The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.

SUMMARY:
The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Tricuspid Regurgitation (TR).

The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.

DETAILED DESCRIPTION:
The main objectives of this study are to evaluate safety and effectiveness of the Mistral implant for the percutaneous treatment of patients with symptomatic moderate or greater tricuspid regurgitation (TR) who are at high risk for tricuspid valve surgery.

Primary endpoints:

* Safety: Incidence of Major Device Related Adverse Events (MDRAE). [Time frame: 6 months].
* Efficacy: Echocardiographic improvement in TR severity of at least 1 grade [Time Frame: 30 days].

Secondary endpoints:

Safety:

* Incidence of Major Device Related Adverse Events (MDRAE). [Time Frame: 1, 6, 12, and 24 months].
* Incidence of device or procedure related serious adverse events [Time Frame: 30 days].

Efficacy:

• Change in TR grade by Echocardiography [Time Frame: 1, 6, 12, and 24 months over baseline].

ELIGIBILITY:
Inclusion Criteria:

* Patient is able and willing to give informed consent, follow protocol procedures, and comply with follow-up visit requirements
* Subject is ≥ 18 years of age or legal age in host country
* Minimum of moderate functional or degenerative tricuspid regurgitation:

  * Subjects with moderate TR: Only NYHA (New York Heart Association) Class III or IV maybe considered for inclusion.
  * Subjects with severe or greater TR: NYHA (New York Heart Association) Class II, III, or IV may be considered for inclusion
* Subject has left ventricular ejection fraction (LVEF) >20 %
* The subject is at high risk of mortality with tricuspid valve surgery as determined by the cardiac surgeon and an interventional cardiologist at the site (center heart team).
* Femoral or Jugular access of the Steerable Catheter with MDS (Mistral Delivery System) is determined to be feasible.
* Subject must agree not to start participating in any other clinical trial for a period of 6 months following the index procedure.
* As determined by the center heart team, the Mistral is the suitable treatment option.

Exclusion Criteria:

* Tricuspid Stenosis >mild
* Tricuspid Sub valvular calcification or calcification of the chordae.
* Subjects with Mitral valve severe stenosis and/or severe regurgitation.
* Previous tricuspid valve repair or replacement that would interfere with placement of Mistral
* Subjects with severe, uncontrolled hypertension.
* Subjects, which need to undergo an emergency surgery.
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoints.
* Subject has a history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 30 days.
* Subject has a history of a myocardial infarction (MI) in the past 30 days.
* Subject has had a percutaneous coronary intervention (PCI), within the last 30 days before procedure.
* Subject with active endocarditis.
* Subject has echocardiographic evidence of intra-cardiac mass, thrombus, vegetation or soft-mobile deposits.
* Subject has hemodynamic instability requiring inotropic or mechanical support.
* Subject has a known hypersensitivity or contraindication to anticoagulant and antiplatelet medication.
* Subject is on chronic dialysis.
* Bleeding disorders or hypercoagulable state.
* In the judgment of the Investigator, co-morbid condition(s) that could limit the subject's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study.
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding.
* Subject has a known allergy to Nitinol alloys, 316L\304 stainless steel.
* Pregnant or lactating women.
* Patients being dependent upon the sponsor or upon the investigator or upon the investigational site.
* According to investigator on site the patient is suffering from a severe end stage disease (e.g. malignancy, severe pulmonary disease, liver disease, renal failure).
* Contraindication for TEE (transesophageal echocardiography) including trans-gastric views.
* Life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
• Safety | 6 months
  Incidence of Major Device Related Adverse Events (MDRAE).

SECONDARY OUTCOMES:
Safety - Incidence of Major Device Related Adverse Events | 1, 6, 12, and 24 months
  Incidence of Major Device Related Adverse Events (MDRAE).
Safety - Incidence of device or procedure related serious adverse events | 30 days
  Incidence of device or procedure related serious adverse events
Effectiveness TR | 1, 6, 12, and 24 months over baseline
  • Change in TR grade by Echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Rubinshtein, Principal Investigator — Wolfson
Locations (1):
- Wolfson Medical Center, Holon, Israel